CLINICAL TRIAL: NCT03851978
Title: Pharmacist Impact on Pneumococcal Polysaccharide Vaccination Rates in Patients With Diabetes in a Supermarket Pharmacy Chain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20014257
Record Dates: First submitted 2019-02-18; First posted 2019-02-22 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Pneumococcal Pneumonia
Keywords: vaccination
MeSH Terms: conditions — Pneumonia, Pneumococcal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist Vaccine Education (Experimental)
  Interventions: Behavioral: Pharmacist Vaccine Education

INTERVENTIONS:
Behavioral: Pharmacist Vaccine Education — When an eligible patient presents to the pharmacy for prescription pick up or drop off, the pop-up note will notify the technician to get a pharmacist for education. The pharmacist will educate the patient on the vaccine and then recommend that the patient receives the vaccine.

SUMMARY:
The goals of the study are to determine the pneumococcal polysaccharide vaccination rate in patients with diabetes before and after community pharmacist education and intervention. Assess barriers of receiving the pneumococcal polysaccharide vaccine in patients with diabetes after pharmacist education in a supermarket chain setting

DETAILED DESCRIPTION:
Three geographically and socioeconomically diverse Kroger pharmacies will be selected in the greater Richmond area. Eligible patients include patients with diabetes between the ages of 19 and 64 and patients who have filled a prescription for at least one diabetes medication in the past 90 days. An NDC (National Drug Code) activity report will be run through Kroger internal reporting to identify patients who have filled a prescription for a diabetes medication in the past 90 days. Excluded patients include those with a known history pneumococcal polysaccharide vaccination, and patients with an allergy to any component of the pneumococcal polysaccharide vaccine. All patients who are deemed eligible will have their immunization history assessed by verifying immunization records in their Kroger medication profile, in the Virginia Immunization Information System (VIIS) or with their primary care physician. The percentage of patients vaccinated with the pneumococcal polysaccharide vaccine in the three Kroger pharmacies will be calculated prior to the start of the intervention period.

Eligible patients will have a pop-up note added to their patient profile in the Kroger system. The pop-up note will indicate that the patient is eligible for education on the pneumococcal polysaccharide vaccine. When an eligible patient presents to the pharmacy for prescription pick up or drop off, the pop-up note will notify the technician to get a pharmacist for education. The pharmacist will educate the patient on the vaccine and then recommend that the patient receives the vaccine. If the patient accepts the recommendation, the pharmacist will then follow Kroger policies and protocol and administer the pneumococcal polysaccharide vaccine to the patient. Standard procedure of administering a pneumococcal vaccine at Kroger includes having the patient complete and sign a vaccination consent form. The consent form consists of questions that assess the patients current health status, immunocompromising conditions, allergies and pregnancy status This indicates to the pharmacist whether the vaccine requested is appropriate for the patient. The pharmacist will review the Kroger consent form and administer the pneumococcal vaccine, using sterile injection technique, if there are no contraindications. After the patient receives the vaccine or declines the vaccine recommendation, the pharmacist will then ask the patient to complete a brief survey. After completion or refusal of the survey, the pharmacist will document the date the survey was completed or denied and if the pneumococcal vaccine was given. After the patient encounter has ended, the pharmacist will edit the pop-up note in the patient profile to document the date the patient was educated, and no further intervention is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes
* Patients who have filled a prescription for at least one diabetes medication in the past 90 days

Exclusion Criteria:

* Patients with a known history pneumococcal polysaccharide vaccination
* Patients with an allergy to any component of the pneumococcal polysaccharide vaccine

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 431 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in vaccination rates | 4 months
  Percentage of patients with diabetes in a national grocery chain pharmacy who received the pneumococcal polysaccharide vaccine before the intervention compared to the percentage who received the vaccination after the intervention.

SECONDARY OUTCOMES:
Barriers to receiving vaccination | 4 months
  Self-reported reasons for not receiving pneumococcal polysaccharide vaccine as measured by a categorical question asking why participants did not receive the vaccine and asking participants to select all reasons that apply and/or provide additional reason(s) not listed.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Venable Goode, Pharm.D., BCPS, FAPhA, FCCP, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - Kroger Pharmacy, Midlothian, Virginia
  - Kroger Pharmacy, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Page A, Harrison A, Nadpara P, Goode JR. Pharmacist impact on pneumococcal polysaccharide vaccination rates in patients with diabetes in a national grocery chain pharmacy. J Am Pharm Assoc (2003). 2020 May-Jun;60(3S):S51-S55.e1. doi: 10.1016/j.japh.2020.02.007. Epub 2020 Mar 17. PMID 32192948